CLINICAL TRIAL: NCT05841641
Title: A Comparative Evaluation of Laser Bandage and Surgical Stent as Palatal Donor Site Dressing After Free Gingival Graft Surgery. A Randomized Control Clinical Trial
Brief Title: Laser Bandage and Surgical Stent as Palatal Donor Site Dressing After Free Gingival Graft Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02_D012_117073
Record Dates: First submitted 2023-02-06; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Palate; Wound
Keywords: LASER BANDAGE; WOUND HEALING
MeSH Terms: conditions — Wounds and Injuries | interventions — Lasers, Semiconductor; Hemostasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser Bandage (Experimental): Graft site charred with Diode Laser at 5 Watts to created charred layer
  Interventions: Device: Laser Bandage
- Hemostatic agent with surgical stent (Experimental): Graft donor site secured with hemostatic agent with surgical stent
  Interventions: Procedure: Hemostatic agent with surgical stent

INTERVENTIONS:
Device: Laser Bandage — The Diode Laser will create a biological bandage at a wavelength of 810 nm, set at 5W in continuous-wave mode, applied via a 400-µm optical fibre.
  Other Names: Diode laser (A.R.C- Fox)
  Arms: Laser Bandage
Procedure: Hemostatic agent with surgical stent — Following graft harvesting, the donor site was secured with a hemostatic agent and protected with a palatal stent
  Other Names: Abgel with surgical stent
  Arms: Hemostatic agent with surgical stent

SUMMARY:
The free gingival graft (FGG) procedure is a harvesting technique that creates an open wound that heals by secondary intention. Retarded wound healing, excessive bleeding, and postoperative pain have been reported after FGG procedures. Hemostatic agents include ferric sub-sulfate solution, absorbable synthetic collagen, absorbable gelatin sponge, or oxidized regenerated cellulose. The agents are often combined with a surgical stent designed to cover the donor site, providing protection and pressure hemostasis. Diode laser also exhibits excellent thermal effects with deep tissue penetrative properties, to enhance coagulation. Laser Bandage (LB) could also enhance wound healing and reduce subjective postoperative complications in the palatal donor area after harvesting FGG similarly.

DETAILED DESCRIPTION:
NEED FOR THE STUDY Autogenous soft tissue grafts are widely used to increase the width of keratinized tissue.1 The free gingival graft (FGG) procedure is a harvesting technique that creates an open wound that heals by secondary intention. Retarded wound healing, excessive bleeding, and postoperative pain have been reported after FGG procedures. To overcome these problems, several techniques and products have been developed. Hemostatic agents such as ferric sub-sulfate solution, absorbable synthetic collagen, absorbable gelatin sponge, or oxidized regenerated cellulose. The agents are often combined with a surgical stent designed to cover the donor site, providing protection and pressure hemostasis. However, these materials may cause adverse effects such as allergies or foreign body reactions or retarded healing of the wound. An optimal method to reduce patient morbidity and enhance early wound healing in the palatal donor site has not yet been defined. Therefore, obtaining new materials that provide better wound care by decreasing bacterial contamination and enhancing wound healing has been considered an essential demand.

Recently, Lasers are also considered a good choice for wound coverage of the donor site due to effective tissue ablation, and hemostatic and bactericidal effects. Laser exhibits hemostatic effects due to its 'hot-tip' effect caused by heat accumulation at the end of the fibre. This produces a thick coagulation layer called a laser bandage or biological bandage. It is also referred to as the 'char layer' or 'eschar on the treated surface. Coleton placed a biological bandage in the donor site using C02 Laser, set at 5W continuous wave in ablative mode. Low and Convissar used erbium laser settings of low wattage with no water, some air and few pulses per second to create laser bandage to achieve coagulation. Since Diode laser also exhibits excellent thermal effects with deep tissue penetrative properties, it enhances coagulation. the investigator proposes Laser Bandage (LB) could also enhance wound healing and reduces subjective postoperative complications in the palatal donor area after harvesting FGG in a similar way.

To date, no studies have evaluated and compared if the diode laser bandage method is more effective than other palatal wound protection methods. Hence, the current study which is first of a kind is undertaken with the objectives of evaluating the effectiveness of Diode LB in achieving donor site hemostasis and comparing wound healing with a standardized palatal haemostatic agent in gel form with the surgical stent in a randomized controlled fashion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing to participate in the study.
2. Patients between the age group of 25 to 55 years.
3. Systemically healthy subjects, non-smokers, no record of allergies
4. Patients with esthetic concerns.
5. Patients with palatal mucosa thickness greater than 4mm
6. Absence of periapical or palatal pathologies and the absence of excessive forces (e.g. mechanical forces from orthodontics and traumatic occlusion).
7. Full mouth plaque score (FMPS) < 20%, Full mouth bleeding score (FMBS) < 20%.

Exclusion Criteria:

1. Patients with any systemic diseases.
2. Patients with a history of coagulation disorders.
3. Patients with immunological disorders.
4. Pregnant and lactating females.
5. History of tobacco usage in any form.
6. Patients taking medication that interfere with healing.
7. Patients with palatal mucosa thickness lesser than 2.5mm.
8. Patients who have undergone periodontal surgery within 6 months from the time they enrolled in the study.

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-12 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
EPITHELIALIZATION | 30 days
  Hydrogen peroxide bubble test

CONTACTS AND LOCATIONS:
Overall Officials: Prabhuji MLV, Principal Investigator — Rajiv Gandhi University of Health Sciences
Locations (1):
- Krishnadevaraya college of dental sciences, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Coleton S. Lasers in surgical periodontics and oral medicine. Dent Clin North Am. 2004 Oct;48(4):937-62, vii. doi: 10.1016/j.cden.2004.05.008. PMID 15464559